CLINICAL TRIAL: NCT00791752
Title: A Randomized, Single-Blind, Placebo-Controlled, Single-Centre, Phase 1Study in Healthy Volunteers to Assess the Safety, Tolerability andPharmacokinetics of AZD4017 After Single Ascending Oral Doses
Brief Title: Study to Investigate Safety and Tolerability Single Ascending Doses of AZD4017
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jan Eriksson MD PhD / Medical Science Director, AstraZeneca R&D Mölndal, Sweden
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: D2060C00001
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: Safety and Tolerability
MeSH Terms: interventions — 2-(1-(5-(cyclohexylcarbamoyl)-6-propylsulfanylpyridin-2-yl)-3-piperidyl)acetic acid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): AZD4017 in ascending doses (start dose 2mg)
  Interventions: Drug: AZD4017
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD4017 — ascending single doses (start dose 2 mg), oral suspension
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The primary aim of this study is to investigate the safety and tolerabilty of AZD4017 when given as single oral ascending doses to healthy volunters. This will be done by comparing the effect of AZD4017 to placebo. The study will aslo investigate the absorption, distrubution and disappearance of AZD4017 in the body. Information about plasma concentrations of AZD4017 vs time after dose intake will also be collected. The future indication for AZD4017 is planned to be Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written and dated informed consent
* BMI between 19 and 30 kg/m2
* Subjects must be willing to use barrier methods of contraception

Exclusion Criteria:

* History of any clinical significant disease
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Laboratory blood sample result showing elevated liverenzymes (ASAT, ALAT) and muscle enzymes (CK).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (Adverse events, vital signs, ECGs, physical examination, laboratoryvariables | The variables will be measure predose and the repeatedly during the following 47 hours after dosing

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax), time to Cmax (tmax), terminal half-life, area under the plasma concentration-time curve and the apparent oral plasma clearance (CL/F) | Blood samples for determination of AZD4017 concenration will be taken predose and repeatedly during the 47 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Hartford, MD PhD, Principal Investigator — Sahlgrenska University Sweden
Locations (1):
- Research Site, Gotteborg, Sweden